CLINICAL TRIAL: NCT00001703
Title: Vaccine Therapy With Tumor Specific Mutated VHL Peptides in Adult Cancer Patients With Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual and lack of peptide vaccine
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Samir N. Khleif, M.D., National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 980139; 98-C-0139 (Other: Clinical Center, NationaI Institutes of Health); 98-C-0139 (Other: Clinical Center, National Institutes of Health); NCT00019526 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2012-06-14 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Renal Cell Carcinoma
Keywords: Immunotherapy; Kidney; Genes; Vaccine Therapy; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — incomplete Freund's adjuvant; montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group A-VHL peptide and ISA-51 adjuvant (Experimental): Patients are vaccinated with 1000 micrograms of the mutant Von Hipple-Lindau (VHL) peptide administered subcutaneously along with ISA-51 adjuvant (Montanide ISA-51 adjuvant, Incomplete Freund's adjuvant) and injected subcutaneously every four weeks for a total of four vaccinations.
  Interventions: Biological: incomplete Freund's adjuvant; Biological: von Hippel-Lindau peptide vaccine

INTERVENTIONS:
Biological: incomplete Freund's adjuvant — 0.7 ml of ISA-51 (Montanide ISA-51 adjuvant, incomplete Freund's adjuvant) will be mixed with peptide alone and injected subcutaneously every four weeks for a total of four vaccinations.
  Other Names: ISA-51; Montanide ISA-51 adjuvant
Biological: von Hippel-Lindau peptide vaccine — 1000 micrograms administered subcutaneously every four weeks for a total of four vaccinations.

SUMMARY:
About 27,000 new cases of renal cell carcinoma (RCC) are diagnosed every year in the United States. 11,000 of these cases will die from the disease. More than half of patients present with advanced or metastatic disease for which chemotherapy plays a very limited role. Therefore, development of another therapeutic approach is needed. Cancers in humans are commonly associated with mutations in dominant and recessive oncogenes. These genes produce mutated proteins that are unique to cancer cells. Von Hipple-Lindau (VHL) gene which is associated with the development of the VHL disease, has been recently mapped and cloned, and it is found to be mutated in 57% of sporadic renal cell carcinomas.

Data in mice have shown the generation of major histocompatibility complex (MHC) restricted cytotoxic T lymphocyte (CTL) that are capable of detecting endogenous cytoplasmic peptide derived from mutated oncogenes. In addition, we have recently demonstrated, by conducting different phase I clinical trials in which we vaccinate cancer patients with mutated Ras or p53 peptides corresponding to the abnormality patients harbor in their tumors, that in some patients we can generate immunological responses represented by the generation of lymphocytes (CD4+ and/or CD8+). In the current study, we would like to extend our observations to test whether VHL tumor suppressor protein can be immunologically targeted by vaccination. We have identified specific epitopes along the amino acid sequence of the VHL protein, which represent known specific human leukocyte antigen (HLA) class-I binding motifs. These amino acids stretches in the VHL protein correspond to the area of the point mutation hot spots. Therefore, we propose to treat patients with sporadic RCC who carry VHL mutations in their tumors with corresponding mutant VHL peptide vaccination. This vaccination will be done either by using pulsed-autologous peripheral mononuclear cells with the peptides, or peptides administered subcutaneously alone or in combination with cytokines.

DETAILED DESCRIPTION:
About 27,000 new cases of renal cell carcinoma (RCC) are diagnosed every year in the United States. 11,000 of these cases will die from the disease. More than half of patients present with advanced or metastatic disease for which chemotherapy plays a very limited role. Therefore, development of another therapeutic approach is needed. Cancers in humans are commonly associated with mutations in dominant and recessive oncogenes. These genes produce mutated proteins that are unique to cancer cells. Von Hipple-Lindau gene, which is associated with the development of the VHL disease, has been recently mapped and cloned; it is found to be mutated in 57% of sporadic renal cell carcinomas.

Data in mice have shown the generation of MHC restricted CTL that are capable of detecting endogenous cytoplasmic peptide derived from mutated oncogenes. In addition, we have recently demonstrated, by conducting different phase I clinical trials in which we vaccinate cancer patients with mutated Ras or p53 peptides corresponding to the abnormality patients harbor in their tumors, that in some patients we can generate immunological responses represented by the generation of lymphocytes (CD4+ and/or CD8+). In the current study, we would like to extend our observations to test whether VHL tumor suppressor protein can be immunologically targeted by vaccination. We have identified specific epitopes along the amino acid sequence of the VHL protein which represent known specific HLA class-I binding motifs. These amino acids stretches in the VHL protein correspond to the area of the point mutation hot spots. Therefore, this protocol treats patients with sporadic RCC who carry VHL mutations in their tumors with corresponding mutant VHL peptide vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older.
* Histologic diagnosis of renal cell carcinoma.
* Tumor tissue availability for determination of Von Hippel-Lindau (VHL) mutation (paraffin block, or fresh tissue).
* Patients must carry a VHL mutation in their tumor.
* Patients must have metastatic disease for which no further chemotherapy or radiation options, which are known to increase survival, are available.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Expected survival more than 3 months.
* While measurable disease is preferable, it is not a necessity.
* The patient should not have received chemotherapy, radiation therapy, immunotherapy or steroids for at least 4 weeks prior to starting vaccination, and should have recovered from all acute toxicities of previous treatment.
* Patients must understand and sign an informed consent document that explains the neoplastic nature of his/her disease, the procedures to be followed, the experimental nature of the treatment, alternative treatments, and potential risks and toxicities.

Exclusion Criteria:

* Any condition that does not fit with the inclusion criteria.
* Any of the following: White blood cells (WBC) less than 2000/mm(3); Platelets less than 100K/mm
* (3); Creatinine greater than 2.0 mg/dl; Serum Bilirubin greater than 2.0 mg/dl, Serum glutamic oxaloacetic transaminase (SGOT), or Serum glutamic pyruvic transaminase (SGPT) greater than 4x normal.
* Human Immunodeficiency virus (HIV) or active Hepatitis B or C (i.e. detectable Hepatitis B surface (HBS) Antigen or Heteroconjugate (HC) antibodies).
* Pregnant women or nursing mothers are ineligible. Women with reproductive potential must have negative urine pregnancy test. Women of reproductive potential must use adequate contraception.
* Patients with active ischemic heart disease (i.e. Class III or IV cardiac disease)-New York Heart Association), a recent history of myocardial infarction (within the last 6 months), history of congestive heart failure, ventricular arrhythmias or other arrhythmias requiring therapy, or any other medical conditions that the principal investigators sees to be unfit for such therapy.
* History of Central Nervous System (CNS) metastases.
* Patients with history of autoimmune disease e.g. (autoimmune neutropenia, thrombocytopenia, or hemolytic anemia; systemic lupus erythematosus, Sjogren syndrome, or scleroderma; myasthenia grave's; Good pasture syndrome; Addison's disease, Hashimoto's thyroiditis, rheumatoid arthritis, multiple sclerosis, or active Graves' disease).
* If, in the opinion of the principal or associate investigators, it is not in the best medical interest of the patient to enter this study, the patient will be ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1998-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir N Khleif, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Cancer Institute, National Institutes of Health, Bethesda, Maryland, United States

REFERENCES:
- [Background] Stahl M, Wilke HJ, Seeber S, Schmoll HJ. Cytokines and cytotoxic agents in renal cell carcinoma: a review. Semin Oncol. 1992 Apr;19(2 Suppl 4):70-9. No abstract available. PMID 1553577
- [Background] Stadler WM, Vogelzang NJ. Low-dose interleukin-2 in the treatment of metastatic renal-cell carcinoma. Semin Oncol. 1995 Feb;22(1):67-73. No abstract available. PMID 7855621
- [Background] Parkinson DR, Sznol M. High-dose interleukin-2 in the therapy of metastatic renal-cell carcinoma. Semin Oncol. 1995 Feb;22(1):61-6. No abstract available. PMID 7855620
- See also: Genetics Home Reference — http://ghr.nlm.nih.gov/
- See also: MedlinePlus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 40-60 total patients may be required for this protocol.
  Between 2-3 years would be required to enter all necessary patients.
Groups:
- Group A-VHL Peptide and ISA-51 Adjuvant: Patients are vaccinated with 1000 micrograms of the mutant Von Hippel-Lindau (VHL) peptide administered subcutaneously along with Montanide ISA-51 adjuvant.
Period: Overall Study
Arm/Group | Group A-VHL Peptide and ISA-51 Adjuvant
Started | 6
Peptide Stock Completed | 3 (off therapy reason for 3 patients)
Completed | 1
Not Completed | 5
Not completed — progressed disease | 2
Not completed — No evidence of disease | 1
Not completed — recurrent disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | Group A-VHL Peptide and ISA-51 Adjuvant
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Generated an Immune Response
Description: The immunological response was assessed by in-vitro T cell cytokine production enzyme-linked immunosorbent spot (ELISPOT). From each patients, post-vaccination peripheral blood mononuclear cells (PBMC) were compared to pre-vaccination as a baseline. A positive ELISPOT result for the patients was defined as a total number of experimental spots in the post-vaccination sample of more than twofold above the total spots in the pre-vaccination sample.
Time Frame: 30 months
Measure: Number; unit: percentage of participants
Arm/Group | Group A-VHL Peptide and ISA-51 Adjuvant
Number analyzed (Participants) | 5
percentage of participants | 80

2. Secondary Outcome: The Number of Participants With Adverse Events.
Description: Here are the total number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 88 months
Measure: Number; unit: participants
Arm/Group | Group A-VHL Peptide and ISA-51 Adjuvant
Number analyzed (Participants) | 5
participants | 5

ADVERSE EVENTS:
Time Frame: 6 1/2 years
Arm/Group | Group A-VHL Peptide and ISA-51 Adjuvant
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A-VHL Peptide and ISA-51 Adjuvant (N=6)
Fatigue (General disorders) | 5 (5)
Injection site reaction (Skin and subcutaneous tissue disorders) | 5 (5)
Headaches (Nervous system disorders) | 4 (4)
myalgia/arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A-VHL Peptide and ISA-51 Adjuvant (N=6)
Fatigue (General disorders) | 5 (5)
Injection site reaction (Skin and subcutaneous tissue disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
Patients were enrolled to Arm A only due to poor accrual and the lack of peptide vaccine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No